CLINICAL TRIAL: NCT00614172
Title: Phase II Trial of Lumpectomy and Partial Breast Proton Therapy for Early Stage Breast Cancer
Brief Title: Proton Therapy for Early Stage Breast Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Loma Linda University (Other)
Responsible Party: Principal Investigator, David Bush, Principal Inverstigator, Loma Linda University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 53294
Record Dates: First submitted 2007-12-26; First posted 2008-02-13 (Estimated); Results first posted 2023-09-21 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2023-08

CONDITIONS: Early-Stage Breast Cancer
Keywords: Proton; Radiation; Breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Protons

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Proton Radiotherapy (Experimental): Two week course of proton radiotherapy to the breast.
  Interventions: Radiation: Proton radiation therapy

INTERVENTIONS:
Radiation: Proton radiation therapy — Proton radiotherapy will start 2-4 weeks following surgical excision. The treatment area will include the lumpectomy site with an additional margin. Daily proton therapy will be given as an out-patient over a two week coarse.

SUMMARY:
The purpose of this study is to determine if partial breast proton therapy is effective treatment for early stage breast cancer following lumpectomy.

DETAILED DESCRIPTION:
Radiation therapy is considered standard treatment for most women with early stage breast cancer following lumpectomy. Post-lumpectomy radiotherapy is a proven treatment that reduces cancer recurrence in the breast and improves survival. When standard whole breast radiation techniques are utilized, portions of the chest wall, lung and heart may also receive significant doses of radiation which can lead to radiation induced complications. Radiation techniques that limit the treatment area to the portion of the breast where the cancer arose can minimize and even eliminate radiation dose to the chest wall, heart and lung. This is called partial breast radiotherapy. This study is designed to evaluate the use of proton beam radiotherapy to deliver partial breast radiotherapy in women with early stage breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* Invasive ductal, medullary, papillary, colloid or tubular histologies
* Stages T1 or T2 (tumors < or = 3 cm) from lumpectomy specimen.
* No more then 3 positive nodes on axillary dissection or negative sentinel node.
* Negative surgical margins (>2mm)

Exclusion Criteria:

* Invasive lobular histology
* Previous chemotherapy for breast cancer
* Extensive intraductal component
* Collagen vascular disease
* Prior malignancy unless disease-free for 5 years
* Patients who are pregnant or lactating

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2004-02; Primary Completion 2020-05-12 (Actual); Study Completion 2020-05-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David A. Bush, MD, Principal Investigator — Loma Linda University Department of Radiation Medicine; Jerry D. Slater, MD, Study Chair — Loma Linda University Department of Radiation Medicine
Locations (1):
- Loma Linda University Medical Center / James M. Slater MD Proton Treatment Center / Department of Radiation Medicine / 11234 Anderson St., Loma Linda, California, United States

REFERENCES:
- [Result] Bush DA, Slater JD, Garberoglio C, Yuh G, Hocko JM, Slater JM. A technique of partial breast irradiation utilizing proton beam radiotherapy: comparison with conformal x-ray therapy. Cancer J. 2007 Mar-Apr;13(2):114-8. doi: 10.1097/PPO.0b013e318046354b. PMID 17476139
- [Result] Bush DA, Slater JD, Garberoglio C, Do S, Lum S, Slater JM. Partial breast irradiation delivered with proton beam: results of a phase II trial. Clin Breast Cancer. 2011 Aug;11(4):241-5. doi: 10.1016/j.clbc.2011.03.023. Epub 2011 Jun 12. PMID 21729673
- [Result] Bush DA, Do S, Lum S, Garberoglio C, Mirshahidi H, Patyal B, Grove R, Slater JD. Partial breast radiation therapy with proton beam: 5-year results with cosmetic outcomes. Int J Radiat Oncol Biol Phys. 2014 Nov 1;90(3):501-5. doi: 10.1016/j.ijrobp.2014.05.1308. Epub 2014 Jul 30. PMID 25084608

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Proton Radiotherapy
Started | 50
Completed | 50
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Females with invasive nonlobular carcinoma greater or less than 3 cm
Groups:
- Partial Breast Radiotherapy With Proton Beam: Two weeks of proton beam radiotherapy to the lumpectomy site
Arm/Group | Partial Breast Radiotherapy With Proton Beam
Number analyzed (Participants) | 50
Age, Continuous [Mean (Full Range); unit: years] | 63 [41 to 83]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 50
  Male | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Histology [Count of Participants; unit: Participants]
  Ductal | 40
  Mucinous | 5
  Tubular | 4
  Medullary | 1
Involved Breast [Count of Participants; unit: Participants]
  Right | 27
  Left | 23
Tumor Size (cm) [Mean (Full Range); unit: CM] | 1.3 [0.3 to 2.8]
ER Receptor Status [Count of Participants; unit: Participants]
  ER+ (>10% Tumor Cells Positive) | 44
  ER- | 6

OUTCOME MEASURES:

1. Primary Outcome: Ipsilateral Breast Tumor Recurrence-free Survival
Description: Lack of tumor recurrence in the treated breast as assessed by imaging and physical exam
Time Frame: Up to 5 years post-treatment completion, average of 48 months
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Partial Breast Radiotherapy With Proton Beam
Number analyzed (Participants) | 50
percentage of patients | 92 [82 to 100]

2. Secondary Outcome: Overall Survival
Description: Overall survival rate at 5 years post-treatment completion.
Time Frame: Up to 5 years post- completion of treatment, average 48 months
Measure: Number (95% Confidence Interval); unit: % Alive
Arm/Group | Partial Breast Radiotherapy With Proton Beam
Number analyzed (Participants) | 50
% Alive | 96 [84 to 100]

ADVERSE EVENTS:
Time Frame: Change between baseline pre-treatment and 5 years post-treatment completion.
Arm/Group | Proton Radiotherapy
All-Cause Mortality (participants affected / at risk) | 2/50
Serious Adverse Events (participants affected / at risk) | 49/50
Other Adverse Events (participants affected / at risk) | 0/50
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Proton Radiotherapy (N=50)
Distant metatastatic disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3)
Isolated axillary occurence (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Events Leading to Death (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) — Metastatic Breast Cancer
Esopageal Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Grade 1 - 2 Acute Skin Toxicity (Skin and subcutaneous tissue disorders) | 30 (30)
Telangiectasia (Blood and lymphatic system disorders) | 13 (13)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2008-04-08): https://cdn.clinicaltrials.gov/large-docs/72/NCT00614172/Prot_SAP_000.pdf